CLINICAL TRIAL: NCT00354172
Title: Transplantation of Umbilical Cord Blood for Myeloid Leukemia Patients Not in CR With Cyclophosphamide/Fludarabine/Total Body Irradiation Myeloablative Preparative Regimen and UCB NK Cells
Brief Title: Donor Umbilical Cord Blood Natural Killer Cells, Aldesleukin and Umbilical Cord Blood Transplant in Patients With Refractory Hematologic Cancers.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing study was started.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMN-2005LS058; MT2005-18 (Other: Blood and Bone Marrow Transplantation Program); 0509M73449 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; previously treated myelodysplastic syndromes; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myeloid, Acute | interventions — aldesleukin; Interleukin-2; Filgrastim; Granulocyte Colony-Stimulating Factor; Therapeutics; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Transplantation, Homologous; Whole-Body Irradiation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated Patients (Experimental): All patients receiving treatment with chemotherapy and radiation, along with natural killer cells, aldesleukin and umbilical cord blood transplant.
  Interventions: Biological: aldesleukin; Biological: filgrastim; Biological: natural killer cell (NK) therapy; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methylprednisolone; Drug: mycophenolate mofetil; Procedure: Umbilical Cord Blood Transplantation (UCBT); Radiation: Total body irradiation (TBI)

INTERVENTIONS:
Biological: aldesleukin — 10 Million units subcutaneous every other day on days -13 (after Natural killer cell graft), -11, -9, -7, -5, -3) If < 45 kilograms (Kg) - interleukin (IL)-2 at 5 MU/m2
  Other Names: IL-2; interleukin-2
Biological: filgrastim — All patients will receive filgrastim (same as granulocyte-colony stimulating factor or G-CSF) 5 mcg/kg/day intravenous (IV) (dose rounded to vial size) based on the actual body weight beginning on day +1 after umbilical cord blood (UCB) infusion. Granulocyte Colony Stimulating Factor (G-CSF) will be administered daily until the absolute neutrophil count (ANC) exceeds 2.5 x 10^9/L for three consecutive days and then discontinued. If the ANC decreases to <1.0 x 10^9/L, G-CSF will be reinstituted.
  Other Names: granulocyte colony-stimulating factor (G-CSF)
Biological: natural killer cell (NK) therapy — All CD3 depleted cells will be given (less those required for product monitoring). The minimum size of a starting NK cell unit will be 700 million mononuclear cells before processing. NK cells (CD56+) and NK cell precursors (CD34+/CD7-, CD34+/CD7+, CD34-/CD7+) will be monitored and reported but will not serve as lot release.
  Other Names: NK cells
Drug: cyclophosphamide — Cyclophosphamide to be administered with high volume fluid flush and mesna on days-18 and -17 after fludarabine. Cyclophosphamide 60 mg/kg/day intravenously (IV) x 2 days, total dose 120 mg/m2 (days -18 and -17)
  Other Names: Cytoxan
Drug: cyclosporine — Patients will receive cyclosporine (CSA) therapy beginning on day -1 maintaining a level of >200 ng/mL. For adults the initial dose will be 2.5 mg/kg intravenously (IV) over 2 hours every 12 hours. For children <40 kg the initial dose will be 2.5 mg/kg IV over 2 hours every 8 hours.
  Other Names: cyclosporin
Drug: fludarabine phosphate — Fludarabine 25 mg/m2/day intravenously (IV) x 3 days, total dose 75 mg/m2 (days -18 to -16)
  Other Names: Fludara
Drug: methylprednisolone — This modification will be enacted based on the engraftment stopping rule on all subsequent patients to stop natural killer (NK) cell reaction.
  Methylprednisolone bolus 1000 mg intravenously (IV) will be administered day -1 and day 0 (before umbilical cord blood transplant) to suppress natural killer (NK) cell activity before transplant. Starting cyclosporin and mycophenolate mofetil (MMF) will also contribute to suppressing residual NK cell activity.
  Other Names: Medrol; Solu-Medrol; Depo-Medrol; methylprednisolone sodium succinate
Drug: mycophenolate mofetil — All patients will begin mycophenolate mofetil (MMF) on day -1. Patients
  ≥ 45 kilograms will receive MMF at the dose of 3 grams/day divided into 2 or 3 doses. Pediatric patient (<45 kilograms) will receive MMF at the dose of 15 mg/kg. Use intravenous (IV) route between days -1 and +5, then, if tolerated, may change to by mouth (PO) between days +6 and +30.
  Stop MMF at day +30 or 7 days after engraftment, whichever day is later, if no acute Graft Versus Host Disease. (Definition of engraftment is 1st day of 3 consecutive days of absolute neutrophil count [ANC] > 0.5 x 10^9 /L).
  Other Names: mycophenolic acid
Procedure: Umbilical Cord Blood Transplantation (UCBT) — The product is infused via intravenous (IV) drip directly into the central line without a needle, pump or filter.
  Other Names: allogeneic transplant
Radiation: Total body irradiation (TBI) — TBI 165 Gray (cGy) will be given twice daily for a total dose of 1320 cGy (days
  -16 to -13).
  Other Names: radiation

SUMMARY:
RATIONALE: Giving chemotherapy, natural killer cells, aldesleukin, and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of abnormal cells and cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine, mycophenolate mofetil, and methylprednisolone before and after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation followed by donor umbilical cord blood natural killer cells, aldesleukin, and umbilical cord blood transplant works in treating patients with refractory hematologic cancer or other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of 6-month disease free survival. The primary laboratory objective is the measure of in vivo expansion of umbilical cord blood (UCB) derived natural killer cells (NK) after a fully ablative preparative regimen.

Secondary

* Determine the incidence of transplant-related mortality at 6 months after NK UCB + double UCBT
* Evaluate the pattern of chimerism after NK UCB + double UCBT
* Determine the incidence of neutrophil engraftment at day 42 after NK UCB + double umbilical cord blood transplantation (UCBT)
* Determine the incidence of platelet engraftment at 6 months after NK UCB + double UCBT
* Determine the incidence of acute graft-versus-host disease (GVHD) grade II-IV and grade III-IV at day 100 after NK UCB + double UCBT
* Determine the incidence of chronic GVHD at 1 year after NK UCB + double UCBT
* Determine the disease-free survival at 1 after NK UCB + double UCBT
* Determine the incidence of relapse at 1 after NK UCB + double UCBT

OUTLINE: This is a single arm, nonrandomized, open-label study.

* Myeloablative conditioning regimen: Patients receive fludarabine intravenously (IV) over 1 hour on days -18 to -16 and cyclophosphamide intravenously (IV) on days -18 and -17. Patients undergo total-body irradiation twice daily on days -16 to -13.
* Haploidentical umbilical cord blood (UCB) natural killer (NK) cell therapy and aldesleukin: Patients undergo haploidentical UCB-enriched NK cell (CD3- depleted) infusion on day -13. Patients then receive aldesleukin subcutaneously on days -13, -11, -9, -7, -5, and -3. Some patients may also receive methylprednisolone IV on days -1 and 0.
* UCB transplantation (UCBT): Patients undergo a single or double UCBT on day 0. Beginning on day 1, patients receive filgrastim (G-CSF) IV once daily until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours 2-3 times daily beginning on day -1 and continuing until day 100, followed by a taper until day 180. Patients also receive mycophenolate mofetil IV or orally 2-3 times daily beginning on day -1 and continuing until day 30 (or 7 days after engraftment) in the absence of acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia with active leukemia (i.e., not in complete remission [CR]), defined by light microscopy (bone marrow) and having failed ≥ 1 round of standard chemotherapy
  * Chronic myelogenous leukemia with myeloid blast crisis not in second chronic phase after ≥ 1 course of standard chemotherapy and imatinib mesylate
  * Myelodysplastic syndromes (MDS) or other myeloproliferative disorders more than 10% blasts after ≥ 1 course of standard chemotherapy
* Unrelated umbilical cord blood (UCB) donor(s) available - Each unit must be 4-6/6 HLA-A, -B, and -DRB1 matched with the recipient (and to each other if 2 units are utilized) (for UCB graft) AND 3/6 HLA-A, -B, and -DRB1 matched with the recipient (for UCB natural killer [NK] cells)
* Karnofsky performance status (PS) 80-100% (adult patients) or Lansky PS 50-100% (pediatric patients)
* Creatinine ≤ 2.0 mg/dL (adult patients) OR creatinine clearance > 40 mL/min (pediatric patients)
* Bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
* Corrected Carbon Monoxide Diffusing Capacity (DLCO) > 50% normal OR oxygen saturation > 92% (in pediatric patients who cannot undergo pulmonary function tests)
* Left ventricular ejection fraction ≥ 45%

Exclusion Criteria:

* Pregnant or nursing
* Positive pregnancy test (Fertile patients must use effective contraception)
* History of HIV infection
* Active infection at time of transplantation

  * Active infection with Aspergillus or other mold within the past 120 days
* Less than 6 months since prior myeloablative transplant (≤ 18 years old)
* Prior myeloablative allotransplant or autologous transplant (> 18 years old)
* No prior extensive therapy including > 12 months of any alkylator chemotherapy or > 6 months of alkylator therapy with extensive radiation (e.g., mantle irradiation for Hodgkin's lymphoma)
* Prior radiation therapy that would make the patient ineligible for total-body irradiation

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated for Refractory Hematologic Cancers: All patients receiving at least partial study treatment with chemotherapy and radiation, along with natural killer cells, aldesleukin and umbilical cord blood transplant.
Period: Overall Study
Arm/Group | Patients Treated for Refractory Hematologic Cancers
Started | 16
Completed | 15 (1 patient did not reach umbilical cord blood transplant)
Not Completed | 1
Not completed — Did not receive transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated for Refractory Hematologic Cancers
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 22 [3 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Patients) Who Were Disease-free and Alive at 6 Months
Description: Number of patients who were alive and free of disease (malignancy) at 6 months after transplant.
Time Frame: 6 Months Post Transplant
Population: One patient did not receive umbilical cord transplant and was not included in this Evaluable patient group.
Measure: Number; unit: Participants
Groups:
- Evaluable Patients: All patients receiving full study treatment with chemotherapy and radiation, along with natural killer cells, aldesleukin and umbilical cord blood transplant.
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 2

2. Secondary Outcome: Number of Participants (Patients) Who Were Disease-free and Alive at 12 Months
Description: Number of patients who were alive and free of disease (malignancy) at 12 months after transplant.
Time Frame: 12 Months Post transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 1

3. Secondary Outcome: Number of Patients Who Were Disease-free and Alive at 24 Months
Description: Number of patients who were alive and free of disease (malignancy) at 24 months after transplant.
Time Frame: 24 Months Post transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 0

4. Secondary Outcome: Number of Participants (Patients) Who Died Due to Transplant.
Description: Patients who had transplant-related mortality (TRM). TRM = adverse event(s) that occur(s) after the patient has received a transplant, the principal investigator decides it is related to the procedure and the patient dies within 6 months.
Time Frame: 6 Months Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 4

5. Secondary Outcome: Number of Participants (Patients) Who Attained Neutrophil Engraftment
Description: Defined as absolute neutrophils (ANC) > 5 x 10^8/Liter for 3 consecutive days.
  ANC is the real number of white blood cells (WBCs) that are neutrophils. The absolute neutrophil count is commonly called the ANC. The ANC is not measured directly. It is derived by multiplying the WBC count times the percent of neutrophils in the differential WBC count. The percent of neutrophils consists of the segmented (fully mature) neutrophils) + the bands (almost mature neutrophils). The normal range for the ANC = 1.5 to 8.0 (1,500 to 8,000/mm3).
Time Frame: Day 42 Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 13

6. Secondary Outcome: Number of Participants (Patients) Who Attained Platelet Engraftment
Description: Platelet engraftment is defined as platelet counts > 50 x 10^9/Liter for 3 consecutive days.
Time Frame: 1 Year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 5

7. Secondary Outcome: Number of Participants (Patients) With Acute Graft-versus-host Disease (GVHD) Grade II-IV
Description: Graft-versus-host disease (GVHD) is a common complication of transplantation in which functional immune cells in the transplanted marrow recognize the recipient as foreign and mount an immunologic attack. The acute or fulminant form of the disease (aGVHD) is normally observed within the first 100 days post-transplant, and is a major challenge to transplants owing to associated morbidity and mortality. Acute GVHD is staged as follows: overall grade (skin-liver-gut) with each organ staged individually from a low of I to a high of IV. Patients with grade IV GVHD usually have a poor prognosis.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 6

8. Secondary Outcome: Number of Participants (Patients) With Acute Graft-versus-Host Disease at Grade III-IV
Description: as for outcome 7
Time Frame: Day 100 post transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 1

9. Secondary Outcome: Number of Participants (Patients) With Chronic Graft-Versus-Host Disease
Description: The chronic form of graft-versus-host-disease (cGVHD) normally occurs after 100 days. The appearance of moderate to severe cases of cGVHD adversely influences long-term survival.
Time Frame: Day 100 through 1 Year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 1

10. Secondary Outcome: Number of Participants (Patients) Who Died by 12 Months
Description: Number of patients who died after receiving treatment within 12 months post transplant.
Time Frame: 1 year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 14

11. Secondary Outcome: Number of Participants (Patients) Who Died by 24 Months
Description: Number of patients who died after receiving treatment within 24 months post transplant.
Time Frame: 2 years post-transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 15

12. Secondary Outcome: Number of Participants (Patients) Who Experienced Relapse by 12 Months
Description: Number of patients who experienced recurrence or progression of disease from the time of transplant.
Time Frame: 1 Year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 10

13. Secondary Outcome: Number of Participants (Patients) Who Experienced Relapse by 24 Months
Description: Number of patients who experienced recurrence or progression of disease from the time of transplant.
Time Frame: 2 Years Post transplant
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 11

14. Secondary Outcome: Number of Participants (Patients) With Successful Natural Killer Cell Expansion
Description: Defined by an absolute circulating donor-derived natural killer cell count of >100 cells/microliter 10-13 days after infusion with <5% donor T and B cells in the mononuclear population
Time Frame: 10-13 Days Post Infusion
Measure: Number; unit: Participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Participants | 3

15. Secondary Outcome: Chimerism After Double Umbilical Cord Blood Transplant (UCBT)
Description: Calculation of Median (range) of percentage of donor cells engrafted (present) in the recipient (patient).
Time Frame: Day 21, Day 100, 6 Months
Population: 1 Year and 2 Year Post Transplant data was not applicable; no patients reached this timeframe to evaluate.
Measure: Median (Full Range); unit: Percentage of Engrafted Cells
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 15
Percentage of Engrafted Cells
  Day 21 | 92 [14 to 100]
  Day 100 | 100 [47 to 100]
  6 Months | 96.5 [93 to 100]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected if deemed related to treatment from Day 1 through 1 year post transplant. It was expected that most treatment related adverse events would occur during this period.
Description: Only serious adverse events were captured for this study.
Arm/Group | Patients Treated for Refractory Hematologic Cancers
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated for Refractory Hematologic Cancers (N=16)
Cardiac failure (Cardiac disorders) | 1 (1)
Death (Blood and lymphatic system disorders) | 4 (4) — Death was due to transplant procedure.
Disease relapse (Blood and lymphatic system disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hemorrhage, lung (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hepatic portal vein flow occluded (Hepatobiliary disorders) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No